CLINICAL TRIAL: NCT03419117
Title: Analgesic Efficacy of Single-shot Erector Spinae Block for Thoracic Surgery
Acronym: AnESTh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jason Wilson, Clinical Instructor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H18-00029
Record Dates: First submitted 2018-01-12; First posted 2018-02-01 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Regional Anesthesia; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Recruited patients will be allocated to an experimental or placebo-control arm. Patients in the experimental arm will receive an ESP block prior to induction of general anesthetic for their thoracoscopic wedge resection, while patients allocated to the placebo-control arm will receive a placebo injection of normal saline in a fashion almost identical to that of the ESP block.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Patients in the experimental arm will receive an ESP block prior to induction of general anesthetic for their thoracoscopic wedge resection
  Interventions: Procedure: ESP block
- Placebo (Placebo Comparator): Patients allocated to the placebo-control arm will receive a placebo injection of normal saline in a fashion almost identical to that of the ESP block.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: ESP block — An ESP block will be performed prior to surgery for postoperative pain control
  Arms: Treatment
Procedure: Placebo — A sham ESP block will be performed before surgery in the placebo group
  Arms: Placebo

SUMMARY:
The erector spinae plane (ESP) block is a novel regional anesthetic technique for the treatment of thoracic, cervical, and abdominal pain. This pilot study aims to investigate the post-operative analgesic effectiveness of ultrasound guided single-shot ESP blocks for patients undergoing minimally invasive thoracoscopic wedge resections of the lung in comparison to those receiving conventional parental opioid analgesia alone. This will be achieved through the use of objective measures including quality the 40 point Quality of Recovery assessment (QoR-40) on postoperative day (POD) 1, visual-analogue pain scale (VAS) in the post-anesthetic care unit (PACU) and at POD 1, and oral morphine-equivalent (OME) opioid consumption in the PACU and at 24 hours post-operatively.

DETAILED DESCRIPTION:
Purpose To investigate the postoperative analgesic effectiveness of the ultrasound-guided ESP block compared to a placebo injection for patients undergoing thoracoscopic wedge resection of the lung.

Hypothesis Thoracoscopic surgery patients who receive an ESP block in addition to current standard of care, consisting of parenteral and enteral opioids and surgical wound infiltration, will have a clinically significant improvement in their QoR-40 at POD 1 and lower pain levels, as measured by VAS in the PACU on arrival and one hour after, and on POD 1, and OME opioid consumption in the PACU and at 24 hours post-operatively, in comparison to those patients who receive the current standard of care along with a placebo injection.

Justification The ESP block is a novel regional anesthetic technique that has shown efficacy in the management of thoracic pain as published in numerous case reports and observational case series. To date, no randomized control trials exist of its efficacy in comparison to conventional parental opioid analgesic management. Thoracoscopic wedge resections of the lung are procedures not usually treated with regional analgesia techniques, but given the moderate pain experienced by many patients, this surgical population will serve as a proof-of-concept for the potential of improved post-operative analgesic and recovery profiles. Proof of analgesic efficacy in this setting may allow a future head-to-head comparison with more invasive analgesic techniques currently used for thoracic surgery such as epidural and paravertebral catheterizations.

In undertaking this aim, we will measure a number of different metrics. The 40-item Quality of Recovery Score (QoR-40) will be our primary objective as it provides a patient-centered global measure of overall health in the postoperative period. It has been tested for validity and reliability, and has undergone quantification for the minimal clinically important difference. Other traditional metrics of analgesic performance including the VAS and 24-hour post-op OME opioid consumption will also be monitored as secondary objectives.

Objectives

Primary Objective:

• Quality-of-Recovery 40 scale at POD 1.

Secondary Objectives:

* Cumulative OME opioid consumption intra-operatively and through PACU, and at 24 hours post operatively.
* Visual analog pain scale assessments post-operatively in PACU on arrival, after 1 hour, and at POD 1.

Research Design The study will be a prospective, single center, randomized, placebo-controlled pilot study requiring 2 patient visits for assessment in the PACU and on POD 1. One interim analysis for safety monitoring will be undertaken.

Sample Size Calculation and Statistical Methods No prior studies have been conducted to calculate an exact sample size calculation. Based on similar work, we will power this study on an expected difference of at least 10 points on the QoR-40 and a SD of 15 when comparing the block to placebo. This is a clinically meaningful difference. Assuming an alpha level of 0.05 and a power of 0.80, our sample size is 74. With a 10% dropout rate we will require recruitment of 82 patients. All outcomes will be analysed with the independent student t-test.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age
* Presenting for elective thoracoscopic wedge resection
* Proficient in the use of the English language
* Able to provide informed consent
* Expected stay > 24 hrs in hospital

Exclusion Criteria:

* ASA greater than, or equal to 4
* Expected post-operative endotracheal intubation
* High likelihood of conversion to open thoracotomy
* A diagnosis of a chronic pain condition
* Depression or other psychiatric diagnosis
* Dementia
* Pregnancy
* Preoperative opioid use >30mg of oral morphine equivalents per day
* Known alcohol or recreational drug abuse
* Contraindication to local anesthetic use including allergy or sensitivity to ropivacaine or other amide-type local anesthetics
* Contraindication to the ESP block or regional anesthetic technique including: allergy or sensitivity to ultrasound gel; previous spine instrumentation; previous rib surgery; injured, diseased, or infected skin overlying the area to be blocked
* Perioperative use, or planned use, of alternative regional anesthetic technique (not including surgical local anesthetic infiltration)
* Perioperative ketamine and lidocaine infusion use

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Quality-of-Recovery 40 (QoR-40) scale at POD 1. | Postoperative day 1. Will be completed on the ward 24hrs after surgery
  The QoR-40 is a widely used and extensively validated measure of quality of recovery

SECONDARY OUTCOMES:
Morphine usage | 30 minutes post-operatively in the PACU and 24hr after surgery.
  Cumulative morphine-equivalent opioid consumption intra-operatively, in PACU (post-anesthetic care unit) and at 24 hours.
Visual analog pain scale (VAS) assessments post-operatively in PACU, and at POD 1. | 30 minutes post-operatively in the PACU and 24hrs after surgery
  Patients will rate their pain on a scale from 0-10 as per standard VAS pain scoring systems.

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Wilson, MD PhD, Principal Investigator — University of British Columbia
Locations (1):
- UBC/Medicine, Faculty of/Anesthesiology, Pharmacology & Therapeutics, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klaibert B, Lohser J, Tang R, Jew M, McGuire A, Wilson J. Efficacy of ultrasound-guided single-injection erector spinae plane block for thoracoscopic wedge resection: a prospective randomized control trial. Reg Anesth Pain Med. 2022 Dec;47(12):749-754. doi: 10.1136/rapm-2022-103602. Epub 2022 Sep 23. PMID 36150741